CLINICAL TRIAL: NCT02069002
Title: Psychosocial Interventions for Indoor Air -Related Functional Symptoms - Randomized Controlled Trial (RCT)
Brief Title: Comparing Interventions for Indoor Air -Related Functional Symptoms
Acronym: TOSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute of Occupational Health (Other)
Collaborators: Finnish Work Environment Fund (Other); The Social Insurance Institution of Finland (Unknown); The Occupational Health Centre of the city of Espoo (Unknown); Terveystalo healthcare service company (Finland) (Unknown); Mehiläinen Oy healthcare service company (Finland) (Unknown); The Occupational Health Centre of the city of Vantaa (Unknown); City of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSR113076; TTL338270202 (Other Grant/Funding Number: Finnish Institute of Occupational Health (Finland))
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2017-02

CONDITIONS: Environmental Illness; Functional Symptoms
Keywords: Indoor Air; Medically unexplained symptoms; Randomized controlled trial; Cognitive-Behavioral Therapy; Applied relaxation
MeSH Terms: conditions — Environmental Illness; Medically Unexplained Symptoms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive-Behavioral Therapy (CBT) (Experimental): There will be ten (10) manualized session, fist 90 minutes and nine (9) 45-minute individual sessions conducted at weekly intervals, last two sessions 2 weeks intervals. One booster session will be conducted three months after the treatment. Sessions include psychoeducation about indoor air related symptoms and personal health behavior factors integrated on patients individual symptomatology, cognitive restructuring, behavioral experiments of patients health promoting behavior, imagery rescripting and relapse prevention.
  Intervention: Behavioral: Psychotherapy (CBT)
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT)
- Applied relaxation group therapy (Experimental): There will be seven (7) manualized session, first 120 minutes and six (6) 90-minute group sessions conducted at weekly intervals, last two sessions 2 weeks intervals. One booster session will be conducted three months after treatment. Sessions include information about indoor air related symptoms, behavioral training and experiments focusing on applied relaxation technique and relapse prevention.
  Intervention: Behavioral: group therapy (ART)
  NB: The Applied Relaxation group Therapy won´t be carried out due to slow and prolonged recruiting process (A steering group agreement 4/2015 and the Ethics Committee approval 5/2015 for the change of the study plan).
  Interventions: Behavioral: Applied relaxation group therapy
- Information session (psychoeducation) (Experimental): There will be one (1) manualized 90-minute individual session. The session includes information about indoor air related symptoms and factors affecting individual health behavior.
  Intervention: Information session (psychoeducation)
  Interventions: Behavioral: Information session (psychoeducation)

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy (CBT)
  Arms: Cognitive-Behavioral Therapy (CBT)
Behavioral: Applied relaxation group therapy
  Arms: Applied relaxation group therapy
Behavioral: Information session (psychoeducation)
  Arms: Information session (psychoeducation)

SUMMARY:
The aim of the current study is to compare the effictiveness of three different psychosocial therapies for treating functional disorders caused by indoor air problems.

DETAILED DESCRIPTION:
Indoor air -related respiratory and other multiple organ symptoms are common in work environments in Finland. Symptoms effect on well-being and quality of life and may lead to impaired social and cognitive functioning and decreased work ability. All indoor air -related conditions are not explained by underlying physical factors and remain medically unexplained. Functional disorders are conditions where patients complain of multiple medically unexplained physical symptoms or physical problems don´t correlate with symptom severity. Indoor air -related symptoms and functional disorders are strongly associated to each other but there are no well-established diagnostic criteria for the condition . So far, there is no available treatment program to the indoor air -related symptoms to offer in primary or occupational health care services in Finland.

In randomized controlled trials, cognitive behavioral treatment has shown to be effective for patients suffering from functional disorders. In addition, a relaxation technique entitled as applied relaxation (Tuomisto & al, 1996) have shown to been shown to been effective to treat different kind of functional problems.

There are no published trials on treatment for individuals of indoor air related symptomatology. The present study is designed as a pragmatic trial to investigate the effect of three different treatment programs as compared to treatment as usual (TAU) for indoor air- related problems in order to improve the (1) work capacity and (2) well-being. A secondary aim of the study is to identify psychological factors affecting the patients' response to the treatment.

The patients are recruited from occupational health care services to establish and to evaluate the efficacy and usability of the treatment procedures. Participants will first undergo baseline assessment including medical examination of the respiratory symptoms. Then they are randomized to one of the study groups: TAU or one of the intervention groups. All study patients receive TAU at occupational health care services for their medical problems during the study. Patients randomized to the study groups receive also the intervention with TAU.

ELIGIBILITY:
Inclusion Criteria:

1. Self-assessed work ability not more than 7 (on a scale 0-10, compared to lifetime best) (removed, see below)
2. Employed minimum three (3) or more years
3. Symptoms related to work environment indoor air (non-industrial workplaces)
4. Respiratory symptoms related to indoor air
5. And symptoms involve more than one other organ system
6. Symptoms onset maximum three years before the study
7. Symptoms are recurrent
8. Symptoms appear more than one (1) environment or continue after repairs environmental exposure(s)
9. No single widely acceptable test of organ system function can explain the symptoms (symptoms are medically unexplained)
10. Minimum of one sick leave due to indoor air symptoms during the preceding half year
11. Fluent Finnish (write/read/speak) (due the interventions)

Exclusion Criteria:

1. six (6) months or more sick leave sick leaves due to indoor air symptoms during the preceding two years and currently unable to work
2. Planned changes in the work (for example retirement, study free period, pregnancy etc.) during the study
3. An acute, untreated medical disorder or illnesses:

   1. Somatic disease that explains the symptoms
   2. An acute, untreated mental disorder (depression, bipolar disorder, psychotic disorders, obsessive-compulsive disorder, eating disorders, personality disorders)
   3. Abuse of narcotics or alcohol or (non-prescribed) medicine
   4. Developmental disorders
4. Psychotherapy (current or has ended preceding two years)
5. No inform consent
6. Other: Patient refusal; not actively participating working life (retired or unemployed)

Based on a steering group´s advice and agreement (10.10.2014), inclusion criteria (Self-assessed work ability not more than 7, on a scale 0-10, compared to lifetime best) was removed. Recruitment continues without this question as an inclusion criteria.

Ages: 25 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-07-29 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
15D - instrument | baseline, 3, 6 and 12 months from the baseline
  The health-related quality of life (HRQoL) instrument (Sintonen, 2001)

SECONDARY OUTCOMES:
• Generalized Anxiety Disorder (GAD-7) | baseline, 3, 6 and 12 months from the baseline
  Self-report measure that assesses anxiety symptoms
Insomnia Severity Index (ISI) | baseline, 3, 6 and 12 months from the baseline
  Self-report measure that assesses insomnia severity
The Symptom checkList-90 (SCL-90) | baseline, 6 and 12 months from the baseline
  Self-report measure that assesses general psychological and somatic symptoms and severity
The Patient Health Questionnaire (PHQ-9) | baseline, 3, 6 and 12 months from the baseline
  Self-report measure that assesses depressive symptoms
Visual Analogue Scale (VAS) | baseline, 3, 6 and 12 months from the baseline
  Self-report measure that assesses respiratory symptom severity
The Acceptance and Action Questionnaire-2 (AAQ-2) | baseline, 3, 6 and 12 months from the baseline
  Self-report measure focuses on experiential avoidance and psychological inflexibility
Illness Worry Scale (IWS) | baseline, 3, 6 and 12 months from the baseline
  Self-report measure that focuses on illness worries and attitudes towards illness
Penn State Worry Questionnaire (PSWQ) | baseline, 3, 6 and 12 months from the baseline
  Self-report measure that focuses on mourning and continuous worrying toughs
Need for Recovery (NRF) | baseline, 3, 6 and 12 months from the baseline
  Self-report measure that focuses on time needed on the recovery after work day
Strategy and Attribution Questionnaire (SAQ) | baseline, 6 and 12 months from the baseline
  Self-report measure focuses on personal attribute strategies.
Self-assessed work ability | baseline, 3, 6 and 12 months from the baseline
  Self-assessed work ability (on a scale 0-10) (Tuomi & al. 1998)

OTHER OUTCOMES:
Working Alliance Inventory (WAI) | after the first, fifth and the last session of the CBT
  Self-report measure that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond; for therapists and the patient of the individual cognitive-behavior therapy
Sense of coherence Group (SOC-G-20) | after the first, fourth and the last session of the grouptherapy
  For the group therapy patients to evaluate the groups therapeutic alliance.
Satisfaction of the treatment | 3, 6 and 12 months from the baseline
  Questionnaire for the intervention groups patients to evaluate the satisfaction of the treatment and its efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Tiina M. Paunio, MD, PhD, Principal Investigator — Finnish Institute of Occupational Health and University of Helsinki
Locations (1):
- Finnish Institute of Occupational Health (Finland), Helsinki, Uusimaa, Finland

REFERENCES:
- [Background] Sintonen H. The 15D instrument of health-related quality of life: properties and applications. Ann Med. 2001 Jul;33(5):328-36. doi: 10.3109/07853890109002086. PMID 11491191
- [Background] Tuomi T Ilmarinen J, Jahkola A, Katajarinne l, Tulkki A (1998) Work ability index. Finnish Institute of Occupational Health, Helsinki.
- [Background] Tuomisto MT, Lappalainen R, Tuomisto T, Timonen T. [Applied relaxation in psychiatry and behavioral therapy]. Duodecim. 1996;112(11):960-7. No abstract available. Finnish. PMID 10592988
- [Derived] Selinheimo S, Vuokko A, Hublin C, Jarnefelt H, Karvala K, Sainio M, Suojalehto H, Paunio T. Psychosocial treatments for employees with non-specific and persistent physical symptoms associated with indoor air: A randomised controlled trial with a one-year follow-up. J Psychosom Res. 2020 Apr;131:109962. doi: 10.1016/j.jpsychores.2020.109962. Epub 2020 Feb 12. PMID 32078837
- [Derived] Selinheimo S, Vuokko A, Hublin C, Jarnefelt H, Karvala K, Sainio M, Suojalehto H, Suvisaari J, Paunio T. Health-related quality among life of employees with persistent nonspecific indoor-air-associated health complaints. J Psychosom Res. 2019 Jul;122:112-120. doi: 10.1016/j.jpsychores.2019.03.181. Epub 2019 Mar 25. PMID 30935665
- [Derived] Selinheimo S, Vuokko A, Sainio M, Karvala K, Suojalehto H, Jarnefelt H, Paunio T. Comparing cognitive-behavioural psychotherapy and psychoeducation for non-specific symptoms associated with indoor air: a randomised control trial protocol. BMJ Open. 2016 Jun 6;6(6):e011003. doi: 10.1136/bmjopen-2015-011003. PMID 27266771
- Available data/document: Study Protocol — http://bmjopen.bmj.com/content/6/6/e011003.full.pdf+html